CLINICAL TRIAL: NCT00104598
Title: Framing Messages for Smoking Cessation With Buproprion
Brief Title: Framing Messages for Smoking Cessation With Bupropion - 6
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Stephanie O'Malley, Director, Division of Substance Abuse Research in Psychiatry, Yale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIDA-13334-6; P50DA013334 (NIH); P50-13334-6
Record Dates: First submitted 2005-03-01; First posted 2005-03-02 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Bupropion

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gain Framed Absitnence Program (Active Comparator): Gain framed video and printed messages encouraging smoking abstinence with Bupropion.
  Interventions: Drug: Bupropion; Behavioral: Smoking Abstinence Program
- Loss Framed Abstinence Program (Active Comparator): Loss framed video and printed messages encouraging smoking abstinence with Bupropion.
  Interventions: Drug: Bupropion; Behavioral: Smoking Abstinence Program

INTERVENTIONS:
Drug: Bupropion
Behavioral: Smoking Abstinence Program — This investigation was a randomized controlled study of two framed message conditions for smoking cessation in combination with open label bupropion SR (300 mg/day). Two hundred fifty-eight cigarette smokers were randomly assigned to receive either gain- or loss-framed video and printed messages encouraging smoking abstinence. Preproduced video and printed information were chosen as the intervention media because of their reliability in delivering specific framed messages. All participants were seen at a community mental health center for 6 months and received a 7-week supply of bupropion SR.

SUMMARY:
This is a randomized study of message framing in individuals beginning a smoking cessation program utilizing bupropion SR and brief counseling, videos, and pamphlets.

ELIGIBILITY:
Exclusion Criteria:

* Pregnant or nursing women, or women of child-bearing potential who are not using an adequate method of contraception
* Psychiatric illnesses requiring psychotropic medications (i.e., psychosis, major depression, mania), or the presence of suicidality or homocidality
* Current use of nicotine replacement therapies (i.e., nicotine patch, gum, or lozenges, nasal spray, or inhaler), bupropion (Zyban, Wellbutrin), or marijuana or current participation in another smoking cessation treatment
* Presence of unstable medical conditions (i.e., cardiac, hepatic, renal disease, diabetes mellitus) that would make a trial of bupropion SR hazardous
* Have taken monoamine oxidase inhibitors or metoprolol succinate within the past six weeks
* History of anorexia nervosa or bulimia
* Previous hypersensitivity to bupropion
* History of alcohol or other drug dependence in the past one year
* History of seizure disorder of any etiology (i.e., brain tumor, traumatic brain injury, substance-induced seizures, etc.)
* Any finding that in the view of the principal investigator would compromise the subject's ability to fulfill the protocol visit schedule and visit requirements or put the subject at risk
* Sharing home or work environment with current or past participant
* No couples or participants who see each other every day

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2000-09; Primary Completion 2004-09 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Smoking Cessation at 7 days | 7-day point prevalence abstinence
Continuous Smoking Abstinence at 6 weeks | 6 weeks
  6-week continuous abstinence.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie O'Malley, Ph.D., Principal Investigator — Substance Abuse Treatment Unit
Locations (1):
- Substance Abuse Treatment Unit, New Haven, Connecticut, United States

REFERENCES:
- [Result] Toll BA, O'Malley SS, Katulak NA, Wu R, Dubin JA, Latimer A, Meandzija B, George TP, Jatlow P, Cooney JL, Salovey P. Comparing gain- and loss-framed messages for smoking cessation with sustained-release bupropion: a randomized controlled trial. Psychol Addict Behav. 2007 Dec;21(4):534-44. doi: 10.1037/0893-164X.21.4.534. PMID 18072836
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961